CLINICAL TRIAL: NCT01692912
Title: A Trial of Active Psoriatic Arthritis (PsA): Randomizing to Treat to a Target vs. Usual Care
Brief Title: Psoriatic Arthritis Treat to Target vs. Usual Care
Acronym: PRC-05-2011
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no enrollment
Sponsor: Pope Research Corporation (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PRC-05-2011
Record Dates: First submitted 2012-09-21; First posted 2012-09-25 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Psoriatic Arthritis (PsA)
Keywords: Psoriatic Arthritis; Randomized; Single blind; Treat to target
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Critical Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive Care (IC) (Active Comparator): Rheumatologists treating to target of DAS28<2.6
  Interventions: Other: Intensive Care
- Routine Care (RC) (No Intervention): Participants treated in the routine manner by their rheumatologist (not treated to the target of DAS28<2.6)

INTERVENTIONS:
Other: Intensive Care — Rheumatologist aims to treat participant in order to achieve a disease activity score improvement of DAS28<2.6
  Arms: Intensive Care (IC)

SUMMARY:
Canadian Rheumatologists will be randomized to treat their participants with active Psoriatic Arthritis to a target (disease activity score <2.6), or as per their routine care. The aim of this study is to determine whether treating to a target results in greater disease improvement than treating patients using routine care.

DETAILED DESCRIPTION:
Canadian Rheumatologists will be randomized to treat their participants with active Psoriatic Arthritis to a target (disease activity score <2.6), or as per their routine care. The aim of this study is to determine whether treating to a target results in greater disease improvement than treating patients using routine care.

ELIGIBILITY:
Inclusion Criteria:

* Psoriatic Arthritis as diagnosed by a rheumatologist and meeting ACR classification criteria for PsA or CASPAR criteria
* The subject must provide written informed consent for participation in the study before any study specific procedures are performed
* Subject has 3 or more SJC on 28 joint count
* Age >=18

Exclusion Criteria:

* Subject has a history of being non-compliant
* Serious concomitant illnesses that in the investigator's opinion negate ability to optimally treat the patient
* If treating with TNF inhibitor, positive PPD > 5mm who have not received INH for recommended course or untreated TB (ie CXR evidence of latent infection). Usual screening is in place for standard of care.
* Pregnancy, breast-feeding or considering pregnancy over the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving low DAS | Month 9 Visit
  The primary outcome measure will be the percentage of patients achieving low Disease Activity Score (DAS<2.6) in each patient group (Intensive Care vs. Routine Care) at the end of the study.

SECONDARY OUTCOMES:
Time to achieving DAS28<2.6 | Month 3 Visit, Month 6 Visit, and Month 9 Visit
  Compares the effectiveness of Intensive Care and Routine Care groups, as measured by the time to achieving target of DAS28<2.6
Absolute change in DAS28 | Month 3 Visit, Month 6 Visit, Month 9 Visit
  To compare the effectiveness of Intensive Care and Routine Care in improving the patient DAS28.
Percentage of Patients achieving ACR 20, 50, and 70 | Month 3 Visit, Month 6 Visit, Month 9 Visit
  ACR 20/50/70 defined as:
  * 20%, 50%, or 70% reduction in tender joint count, and
  * 20%, 50%, or 70% reduction in swollen joint count, and
  * a 20%, 50%, or 70% reduction in 3 of the following 5 measures:
  * Patient and physician global assessments (VAS)
  * Patient pain score (VAS)
  * HAQ-DI
  * ESR or CRP
Percentage of patients achieving PsARC | Month 3 Visit, Month 6 Visit, Month 9 Visit
  PsARC defined as improvement in at least 2 of the 4 following measures, one of which must be joint swelling or tenderness, and no worsening in any of the 4 measures:
  * MDGA (0-5 point scale): reduction by 1 point.
  * PGA (0-5 point scale): reduction by 1 point.
  * TJC (76 or 68): reduction by >=30%.
  * SJC (76 or 68): reduction by >=30%.
Absolute change in HAQ-DI | Month 3 Visit, Month 6 Visit, Month 9 Visit
  HAQ-DI is a self-administered questionnaire using the patient's functional ability during the last week. It consists of 20 items converging to 8 scales measuring dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. The patients rate each activity as 0 = without any difficulty, 1 = some difficulty, 2 = much difficulty and 4 = unable. The final score ranges from 0 to 3 with higher scores indicating more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Janet E. Pope, MD, MPH, FRCPC, Principal Investigator — Pope Research Corp., University of Western Ontario, St. Joseph's Health Care London
Locations (4):
- Canada (4):
  - Pope Research Corp., 68 Green Acres Drive, London, Ontario
  - The Arthritis Program Research Group, Newmarket, Ontario
  - Arthur Karasik, Toronto, Ontario
  - Institut de Rheumatologie de Montreal, Montreal, Quebec